CLINICAL TRIAL: NCT00582491
Title: Modafinil, Sleep, and Cognition in Cocaine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 0607001659; R01DA011744 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Cocaine Dependence; Substance-induced Sleep Disorder; Substance-induced Cognitive Disorder
Keywords: Modafinil; Sleep; Cognition; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Modafinil 400mg orally everyday for 16 days
  Interventions: Drug: Modafinil
- II (Placebo Comparator): Placebo orally everyday for 16 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — Modafinil 400mg orally every day for 16 days
  Other Names: Provigil
  Arms: I
Drug: Placebo — Placebo orally everyday for 16 days
  Arms: II

SUMMARY:
Subjects participating in this protocol will participate in three phases: 1) pre-admission, 2) inpatient admission, and 3) follow-up. Pre-admission involves screening (detailed in inclusion/exclusion criteria section) and one week of outpatient sleep and activity monitoring. Inpatient admission is 16 consecutive nights on the Clinical Neuroscience Research Unit and involves subjective and objective tests of sleep, sleepiness, attention, and learning. During inpatient admission subjects will take modafinil or placebo. For follow-up, subjects will return to the CNRU for one night and again participate in objective tests of sleep, sleepiness, attention, and learning. We hypothesize that modafinil will decrease subject and objective measures of sleepiness and will promote attention and learning in cocaine dependent persons.

DETAILED DESCRIPTION:
A relatively new treatment for the excessive daytime sleepiness (EDS) associated with inadequate sleep is the drug modafinil. Modafinil decreases subjective reports and objective measures of daytime sleepiness under conditions of sleep restriction, while enhancing cognitive performance. At the same time, sleep quality does not appear to be affected significantly. Interestingly, recent clinical trials in cocaine-dependent populations suggest that modafinil reduces the relapse to cocaine use, by unknown mechanisms.

We propose to employ both subjective and objective measures of nocturnal sleep and daytime sleepiness, as well as measures of general cognitive performance and sleep-dependent memory consolidation, to explore potential mechanistic relationships between cocaine abstinence, EDS, and modafinil's efficacy in preventing cocaine relapse.

The following specific aims are proposed:

Specific Aim 1: To establish whether objective measures of poor nocturnal sleep (e.g., reduced total sleep time and sleep efficiency) that progressively characterize periods of sustained cocaine abstinence are also associated with objective evidence of excessive daytime sleepiness (EDS).

Specific Aim 2: To establish the ability of modafinil to reverse the excessive daytime sleepiness (EDS) and deficits in cognitive performance that characterize cocaine abstinence.

Specific Aim 3: To conduct a pilot study to determine whether the observed abnormalities in objective sleep, EDS, and/or cognitive function predict relapse to cocaine use and/or whether successful abstinence from cocaine is associated with normalization of the same.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals, ages 18-65, meeting current DSM-IV criteria for cocaine dependence. Documented positive urine toxicology screen for cocaine at intake and regular 3 times more weekly use of cocaine.
* Subject has voluntarily given informed consent and signed the informed consent document(s).
* Able to read English and complete study evaluations.

Exclusion Criteria:

* Use of prescription medication in the past 6 months indicating a medical or psychiatric condition that in the opinion of the PI would interfere with study participation (e.g. hypertension, severe renal or hepatic disease, HIV, primary psychotic disorder, primary mood disorder, primary sleep disorder).
* Meeting DSM-IV criteria for dependence on any substance other than cocaine and nicotine.
* Significant underlying medical or psychiatric conditions or hypersensitivity to modafinil that in the opinion of the PI would interfere with study participation.
* Abstinence from cocaine for more than one week prior to inpatient admission.
* Positive urine or serum pregnancy test.
* Women who are pregnant or lactating, or not using a reliable method of birth control.
* (For subjects completing the fMRI portion of the study) Presence of or history indicative of ferromagnetic metal in their bodies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Morgan, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 participants with self-identified cocaine problems responded to newspaper advertisements and passed initial telephone screening. Of those who passed the telephone screening, 29 were found to be qualified for participation after in-person screening. 21 participants entered the study and were subsequently randomized.
Groups:
- Modafinil 400mg: Modafinil 400mg orally everyday for 16 days
Period: Overall Study
Arm/Group | Modafinil 400mg | Placebo
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Modafinil (400mg): Participants received single oral dose of modafinil (400mg) every morning for 16 days
- Placebo: Participants received a single oral placebo every morning for 16 days
- Total: Total of all reporting groups
Arm/Group | Modafinil (400mg) | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 41.9 (3.7) | 43.9 (8.4) | 42.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time (Minutes)
Description: Total sleep time was defined as the time from sleep onset until final awakening minus the time awake after sleep onset.
  Experimental polysomnographic sleep measurement was performed on the following three study night blocks: 1 to 3, 7 to 9, and 14 to 16. Data from each three-night block were averaged and reported as weeks 1, 2, and 3 respectively.
Time Frame: After 1 Week
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Minutes | 364 (75) | 379 (38)

2. Secondary Outcome: Overall Sleep Quality on Visual Analog Scale (Millimeters)
Description: Upon awakening, participants rated their "overall quality of sleep". Ratings were indicated by the participants marking an "X" on 100 mm lines (ie "worse," "best"). The placement of the "X" was measured, using a ruler, to the nearest millimeter and thus ranged from 0 mm to 100 mm. Lower scores correspond to a worse quality of sleep and higher scores correspond to a better sleep quality.
  Subjective measures from days 1 to 3, 7 to 9, and 14 to 16 were averaged to correspond to weeks 1, 2, and 3.
Time Frame: After 1 Week
Population: The number of participants who completed the study were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Millimeters | 63 (21) | 59 (23)

3. Primary Outcome: Total Sleep Time (Minutes)
Description: as for outcome 1
Time Frame: After 2 Weeks
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Minutes | 383 (40) | 343 (45)

4. Primary Outcome: Total Sleep Time (Minutes)
Description: as for outcome 1
Time Frame: After 3 Weeks
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Minutes | 373 (42) | 315 (51)

5. Primary Outcome: Time Spent in Sleep Stage 3 (Minutes)
Description: Experimental polysomnographic sleep measurement was performed on the following three study night blocks: 1 to 3, 7 to 9, and 14 to 16. Data from each three-night block were averaged and reported as weeks 1, 2, and 3 respectively.
Time Frame: After 1 Week
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Minutes | 73 (33) | 36 (33)

6. Primary Outcome: Time Spent in Sleep Stage 3 (Minutes)
Description: as for outcome 5
Time Frame: After 2 Weeks
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Minutes | 83 (29) | 36 (26)

7. Primary Outcome: Time Spent in Sleep Stage 3 (Minutes)
Description: as for outcome 5
Time Frame: After 3 Weeks
Population: The number of participants who completed the study were analyzed
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Minutes | 92 (27) | 44 (31)

8. Secondary Outcome: Overall Sleep Quality on Visual Analog Scale (Millimeters)
Description: as for outcome 2
Time Frame: After 2 Weeks
Population: The number of participants who completed the study were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Millimeters | 79 (16) | 70 (18)

9. Secondary Outcome: Overall Sleep Quality on Visual Analog Scale (Millimeters)
Description: as for outcome 2
Time Frame: After 3 Weeks
Population: The number of participants who completed the study were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Modafinil (400mg) | Placebo
Number analyzed (Participants) | 10 | 10
Millimeters | 81 (20) | 75 (16)

ADVERSE EVENTS:
Time Frame: Throughout the length of the study (approximately 2 1/2 years)
Arm/Group | Modafinil (400mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Modafinil (400mg) (N=10) | Placebo (N=10)
Back/Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 1
Heart Palpitations (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes